CLINICAL TRIAL: NCT04128722
Title: TOPical Sirolimus in linGUal Microcystic Lymphatic Malformation -TOPGUN
Acronym: TOPGUN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DR190041-TOPGUN; 2019-001530-33 (EudraCT Number)
Record Dates: First submitted 2019-09-24; First posted 2019-10-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lingual Microcystic Lymphatic Malformations
Keywords: LMLM; Sirolimus

STUDY DESIGN:
Intervention Model Description: Individually randomized stepped wedge
Who Masked: Outcomes Assessor
Masking Description: Primary outcome is assessed on anonymised photographs by an adjudication committee blinded from treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus 1mg/mL (Experimental): Application of 1 mg/mL sirolimus solution, 0.5 mL to 1 mL according to the size of the lesion, once daily, on lingual microcystic lymphatic malformation, the experimental intervention versus usual care (no treatment), the control condition.
  Interventions: Drug: Sirolimus Oral Liquid Product 1mg/mL
- Control condition (No Intervention): Usual care, i.e. no intervention

INTERVENTIONS:
Drug: Sirolimus Oral Liquid Product 1mg/mL — 0.5 mL to 1 mL according to the size of the lesion, once daily, on lingual microcystic lymphatic malformation
  Other Names: Experimental treatment
  Arms: Sirolimus 1mg/mL

SUMMARY:
Lingual microcystic lymphatic malformations (LMLMs) are rare congenital vascular malformations, presenting as clusters of cysts filled with lymph fluid or blood. They are responsible for a heavy burden even with small well-limited lesions because of oozing, bleeding, infections, or even speech, chewing or breathing impairment. Pain and aesthetic prejudice are also frequently reported. The natural history of LMLMs is progressive worsening. LMLMs complex management requires multidisciplinary care in specialised centres, and the "wait-and-see" approach is frequently used. In complicated lymphatic malformations, whatever the location, treatment with oral sirolimus, an mTOR (mammalian Target of Rapamycin) inhibitor, is often used.

Topical sirolimus is a known effective treatment for some cutaneous conditions such as angiofibromas in tuberous sclerosis. Topical applications of sirolimus on the buccal mucosae have been reported in erosive lichen planus and oral pemphigus vulgaris with good tolerance and none to slight detectable blood sirolimus concentrations.

The objective of this study is to evaluate the efficacy and safety of a 1mg/mL sirolimus solution applied once daily on mild to moderate lingual microcystic lymphatic malformation in children and adults after 4, 8, 12, 16, 20 and 24 weeks of treatment as compared to usual care (no treatment).

DETAILED DESCRIPTION:
This is a randomized, open-labelled, multicenter pilot study using an individually randomized stepped wedge design over a 24 weeks period to evaluate topical application of 1 mg/mL sirolimus solution, 0.5 mL to 1 mL according to the size of the lesion, once daily, on lingual microcystic lymphatic malformation that do not require systemic treatment, the experimental intervention versus usual care (no treatment), the control condition.

In this design, subjects are included in a cohort where at a randomized time (W0, W4, W8 or W12), they switch from an observational period to the interventional period.

All subjects will be followed for 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 5 years of age
* Lingual microcystic lymphatic malformation that does not require systemic treatment, assessed by clinical examination and head-and-neck MRI imaging prior to study enrolment, with or without underlying syndromic malformation (CLAPO for instance)
* Participants covered by or having the rights to social security
* Written informed consent obtained from participant and participant's legal representative if participant is under 18
* Ability for participant to comply with the requirements of the study

Exclusion Criteria:

* Patients with a lymphatic malformation requiring a continued background therapy (involving deep organs)
* Secondary lymphatic malformations (lymphangiectasia post-radiotherapy, etc)
* Previous treatment with systemic or topical mTOR (mammilian target of rapamycin) inhibitors within 12 months before inclusion (half-life of oral sirolimus is 60 days in adults).
* Previous treatment with oral or topical steroids within 10 days before inclusion (half-life of corticosteroids is 12-36 hours)
* Immunosuppression (immunosuppressive disease or immunosuppressive treatment)
* Ongoing neoplasia
* Active chronic infectious disease (Hepatitis-B virus, Hepatitis-C virus, HIV, etc)
* Local necrosis
* Local fungal, viral (herpes simplex virus, varicella zoster virus, etc) or bacterial infection on the site of the LMLM (based on clinical examination)
* Known allergy to one of the components of the sirolimus solution
* Soy bean or Peanut allergy
* Pregnant or breastfeeding women
* Women of child-bearing potential (including teenagers) not using a reliable contraceptive method until the end of the study and three month after the end of the study or sirolimus discontinuation.
* Already involved in another therapeutic trial

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Change in Physical Global Assessment (PGA) after topical application of Sirolimus for 12 weeks | 12 weeks
  The primary outcome will consist in the evaluation of global severity of the LMLM using PGA (Physical Global Assessment) 0 to 5 score, by three independent blinded experts, on monthly standardized photographs.
  A 1-point improvement versus baseline in PGA scale would already have a clinical relevance.
  Our primary analysis will focus on change in PGA after topical application of Sirolimus for 12 weeks

SECONDARY OUTCOMES:
Investigator-assessed PGA | at weeks 0, 4, 8, 12, 16, 20 and 24
  Investigator-assessed PGA (Physical Global Assessment)
Assessment by the patient regarding severity of oozing, bleeding, sialorrhea, eating impairment, taste modification, aesthetic impairment, pain and global discomfort, | at weeks 0, 4, 8, 12, 16, 20 and 24.
  Assessment by the patient regarding severity of oozing, bleeding, sialorrhea, eating impairment, taste modification, aesthetic impairment, pain and global discomfort, each using a numeric scale from 0 to 10 (0: clear, 10: very severe), at weeks 0, 4, 8, 12, 16, 20 and 24
Global evolution assessed by the patient | at weeks 4, 8, 12, 16, 20 and 24.
  Global evolution assessed by the patient from -10 to 10 (-10 = severe worsening, 0 = no change, 10 = complete recovery), at weeks 4, 8, 12, 16, 20 and 24.
Global Quality of life assessment | at baseline, at time of switch to the intervention (either week 0, week 4, week 8 or week 12) and week 24.
  (DLQI or children's DLQI for minors aged 5 to 16), at baseline, time of switch to treatment and week 24.
Measurements of the lesion | at baseline, at time of switch to the intervention (either week 0, week 4, week 8 or week 12) and week 24.
  by the investigator, at baseline, time of switch to treatment and week 24.
Time to obtain optimal results | up to 24 weeks
  i.e. time from switch to treatment to time reaching the minimal PGA score
Assessment of tolerance of topical sirolimus: | from the switch to intervention up to the end of the study, i.e a maximum of 24 weeks.
  record of local side effects at each visit after the patient has crossed over to the intervention, up to 24 weeks
General side effects | rom the switch to intervention up to the end of the study, i.e a maximum of 24 weeks.
  Follow-up of general side effects
Assessment of sirolimus blood passage | after 4 weeks of treatment, then 8 weeks, then every 8 weeks until week 24
  by measuring residual sirolimus blood concentration: after 4 weeks of treatment, then 8 weeks, then every 8 weeks until week 24
Evaluation of biological safety | after 8,16 and up to 24 weeks
  Number of participants with at least one biological abnormality treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Annabel MARUANI, MD-PhD, Study Director — University Hospital of TOURS;INSERM 1246 SPHERE
Locations (2):
- France (2):
  - Univsersity of TOURS _ Service de Dermatologie, Tours, Indre et Loire
  - Hospital NECKER -AP-HP - Dermatology, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marchand A, Caille A, Gissot V, Giraudeau B, Lengelle C, Bourgoin H, Largeau B, Leducq S, Maruani A. Topical sirolimus solution for lingual microcystic lymphatic malformations in children and adults (TOPGUN): study protocol for a multicenter, randomized, assessor-blinded, controlled, stepped-wedge clinical trial. Trials. 2022 Jul 8;23(1):557. doi: 10.1186/s13063-022-06365-y. PMID 35804404